CLINICAL TRIAL: NCT03863262
Title: Screening for Depression in cADiovasCular pAtients at a Tertiary Center in Trinidad.
Acronym: SAD-CAT
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Other Study IDs: CEC691/08/18
Record Dates: First submitted 2019-02-20; First posted 2019-03-05 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: cardiovascular
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This was an observational study aimed to screen patients with cardiovascular disease for depression in Trinidad and Tobago in a tertiary center and to determine if there is a significant association between patients with symptoms of depression and other comorbidities. Patients (N=1203) were randomly selected from the outpatient cardiology clinics at the Eric Williams Medical Sciences Complex. After fulfilling the inclusion criteria and informed consent were obtained, they were given the case report form which included the Patient Health Questionnaire 9.

DETAILED DESCRIPTION:
The study design was a cross-sectional descriptive study performed from November 2018 to February 2019. It was performed at the Eric Williams Medical Sciences Complex, Champ Fleurs, Trinidad. The primary objectives of the study were to screen patients for depression in those with cardiovascular disease in Trinidad and Tobago and to determine the association between patients with depression and other comorbidities.

Patients were targeted for participation in the study while waiting to see the attached physician to the cardiology clinic. Participants were attained at the Eric Williams Medical Sciences Complex during the days Monday to Friday where there were ongoing cardiology outpatient clinics. Once informed consent was obtained from these patients, a questionnaire was administered to these patients in which the primary investigator and/or co-investigator was/were present on site. The number of participants in this study was 1203 patients. There were no dropped subjects from the study nor were there any incomplete questionnaires by any participants. The sample size for this study was calculated to be 1159 patients. Based on a study done by Huffman, it was estimated that 40% of patients with cardiovascular disease also have depression(2). The Type I error rate 5% (α = 0.05) making the Type II error rate 95% (β = 0.95) with a statistical power of 90%. Assuming a 10% patient decline and attrition rate and a minimum detectable difference of 10%, the estimated sample size was calculated to be 1159 patients.

Data collection was performed by the researchers of the study along with eight specifically trained and oriented medical students. All data collectors in the study were supervised by primary investigator and co-investigator of the study so that in the event of any adverse events such as acute psychosis or any acute cardiology emergencies, patients could have been referred directly to the accident and emergency department at Eric Williams Medical Sciences Complex where routine medical care could have been executed.

Additionally, there was an attached consent form which was also approved by the ethical committee of the University of the West Indies, St. Augustine. This consent form clearly explained to the participants why the research was being conducted, the average duration of completing the questionnaire, the benefits and any potential risks associated with participation in the study along with the assurance that confidentiality will be maintained throughout the entire study and that the patient can stop or not complete the questionnaire at any point without any facing repercussions. This information was documented on the consent form and also explained by the researchers of the study to each potential participant. All additional questions from patients were answered truthfully regardless of if it would have affected the patient's decision to participate in the study.

Patients were asked to participate in the study as long as they were registered patients at Eric Williams Medical Sciences Complex in any of the cardiology outpatient clinics. This was confirmed by matching patients with their registration numbers on the cardiology outpatient clinic appointment listings. These lists are made prior to each cardiology clinic that is scheduled every week on Mondays, Tuesdays, Wednesdays, Thursdays and Fridays. The inclusion criteria for participation in the study included patients who were 18 years old and over along with registered patients of the cardiology outpatient clinics at Eric Williams Sciences Complex.

Of note, no rewards or incentives were offered to encourage participation in the study by subjects nor were there any penalization for declining participation in the study. Specifically, patients were not offered any monetary payments to encourage their participation in the study. Patients were allowed to decide on their own, whether or not they wanted to participate in the study. Subjects were able to participate based on the fulfilling inclusion criteria and informed consent attained. Of significance, there was no sponsorship obtained to conduct this study.

Confidentiality of patients was kept and ensured as no patient names were recorded and all data recorded was de-identified. Patients were uniquely identified using their clinic registration numbers of the cardiology outpatient clinic. By using registration numbers to identify patients, this assisted in preventing duplicate collection and entry of data. Additionally, the database was only accessible to the primary investigator and the co-investigator of the study. The data was stored on a device which was password protected and again this password was only available to the primary investigator and co-investigator of the study. The database was encrypted to ensure the patient's recorded information was safe.

Of importance, no invasive data was collected from participants in this study. No blood samples were drawn and no drugs being tested were administered to any patients enrolled in the study. Additionally, any patients deemed as medical emergencies had the opportunity to be referred to the accident and emergency department of Eric Williams Medical Sciences Complex where the routine medical protocol was followed and appropriate referrals were made. Some examples of these emergencies included acute psychosis, acute coronary syndromes, and acute heart failure.

The scores of the Patient Health Questionnaire-9 were verbally communicated to the patients in confidentiality by the primary investigator and or co-investigator of the study along with the interpretation of the score and what it meant on the depression scale. Patients were given the opportunity to decide if they wanted these results communicated to the physician seeing them in the cardiology outpatient clinic and if so; the results were given to their respective physicians who would have decided on appropriate referrals and routine medical care. This would include appropriate referrals to psychiatry.

The Social Sciences 24 (SPSS, Chicago, Illinois USA) was the software used for the entry of data and its analysis. Descriptive analyses were performed which were unadjusted. Statistical significance was accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Registered patients at Eric Williams Medical Sciences Complex in any of the cardiology outpatient clinics. This was confirmed by matching patients with their registration numbers on the cardiology outpatient clinic appointment listings. These lists are made prior to each cardiology clinic that is scheduled every week on Mondays, Tuesdays, Wednesdays, Thursdays and Fridays.
* Patients who were 18 years old

Exclusion Criteria:

* Patients less than 18 years old
* Those who did not give informed consent to participate in the study
* Patients who were not registered patients of the cardiology outpatient clinics at Eric Williams Medical Sciences Complex along
* Patients who were acutely unwell requiring hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The number of participants in this study was 1203 patients. There were no dropped subjects from the study nor were there any incomplete questionnaires by any participants. The sample size for this study was calculated to be 1159 patients.
  Based on a study done by Huffman, it was estimated that 40% of patients with cardiovascular disease also have depression(2). The Type I error rate 5% (α = 0.05) making the Type II error rate 95% (β = 0.95) with a statistical power of 90%. Assuming a 10% patient decline and attrition rate and a minimum detectable difference of 10%, the estimated sample size was calculated to be 1159 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1203 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of cardiovascular patients with a PHQ9 Score > 10 | 4 months
  The percentage of cardiovascular patients with a screening for depression score > 10.

SECONDARY OUTCOMES:
Demographic associations with a PHQ9 Score >10. | 4 months
  Demographic associations with respect to a PHQ Score >10

CONTACTS AND LOCATIONS:
Locations (2):
- Trinidad and Tobago (2):
  - Eric Williams Medical Sciences Complex, Port of Spain, North
  - The University of the West Indies, Saint Augustine, North

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huffman JC, Celano CM, Beach SR, Motiwala SR, Januzzi JL. Depression and cardiac disease: epidemiology, mechanisms, and diagnosis. Cardiovasc Psychiatry Neurol. 2013;2013:695925. doi: 10.1155/2013/695925. Epub 2013 Apr 7. PMID 23653854
- [Result] Zellweger MJ, Osterwalder RH, Langewitz W, Pfisterer ME. Coronary artery disease and depression. Eur Heart J. 2004 Jan;25(1):3-9. doi: 10.1016/j.ehj.2003.09.009. PMID 14683736
- [Result] Whooley MA. Depression and cardiovascular disease: healing the broken-hearted. JAMA. 2006 Jun 28;295(24):2874-81. doi: 10.1001/jama.295.24.2874. PMID 16804154
- [Result] Wittkampf K, van Ravesteijn H, Baas K, van de Hoogen H, Schene A, Bindels P, Lucassen P, van de Lisdonk E, van Weert H. The accuracy of Patient Health Questionnaire-9 in detecting depression and measuring depression severity in high-risk groups in primary care. Gen Hosp Psychiatry. 2009 Sep-Oct;31(5):451-9. doi: 10.1016/j.genhosppsych.2009.06.001. Epub 2009 Jul 10. PMID 19703639
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Seecheran N, Jagdeo CL, Seecheran R, Seecheran V, Persad S, Peram L, Evans M, Edwards J, Thackoorcharan S, Davis B, Davis S, Dawkins B, Dayaram A, De Freitas M, Deonarinesingh T, Dhanai J, Didier C, Motilal S, Baboolal N. Screening for depressive symptoms in cardiovascular patients at a tertiary centre in Trinidad and Tobago: investigation of correlates in the SAD CAT study. BMC Psychiatry. 2020 Oct 8;20(1):498. doi: 10.1186/s12888-020-02909-1. PMID 33032571

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03863262/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03863262/ICF_001.pdf